CLINICAL TRIAL: NCT03050034
Title: Role of Wireless Monitoring in Internal Medicine Unit for Ongoing Assessment of Acute Instable Patients: Impact on Outcomes, Length of Stay and Costs.
Brief Title: Role of Wireless Monitoring in Internal Medicine Unit for Ongoing Assessment of Acute Instable Patients
Acronym: LiMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Socio Sanitaria Territoriale del Garda (Other Government)
Collaborators: ASST-Garda: Internal Medicina Unit Manerbio Hospital (BS) (Unknown); University of Modena and Reggio Emilia (Other); Milano-Bicocca University Medical Statistic Department (Unknown)
Responsible Party: Principal Investigator, Filomena Pietrantonio, Internal Medicin Unit Director, Azienda Socio Sanitaria Territoriale del Garda
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIMS2017
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Wireless Vital Signs Monitoring System; Acutely Ill Complex and Poly-pathological Patients; Internal Medicine Unit Mission
Keywords: Wireless monitoring system; Acute Medicine; Poly-pathological patients; Internal Medicine core competencies; Acute Complex Care Model

STUDY DESIGN:
Intervention Model Description: Pilot perspective controlled randomized open-label single-center study to evaluate the management of critically ill patients hospitalized comparing vital signs wireless monitoring versus conventional monitoring in the first 72 h of hospitalization extendable to 5 days if the MEWS after 72 h is even greater than or equal to 3 and/or the NEWS is greater than or equal to 5.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vital signs wireless monitoring system (Experimental): All patients with MEWS (Modified Early Warning Score) greater than or equal to 3 and/or NEWS (National Early Warning Score) greater than or equal to 5, at admission, regardless of the reason for hospitalization and all patients with glycemic decompensation and/or severe fluid and electrolyte imbalance, regardless of MEWS/ NEWS, undergone to continuous monitoring with wireless monitoring system WIN @ Hospital.
  Interventions: Device: WIN @ Hospital system
- Control arm (Active Comparator): All patients with MEWS (Modified Early Warning Score) greater than or equal to 3 and/or NEWS (National Early Warning Score) greater than or equal to 5, at admission, regardless of the reason for admission and all patients with glycemic decompensation and/or severe fluid and electrolyte imbalance, regardless of MEWS NEWS undergone to traditional monitoring performed at regular intervals by the nursing staff.
  Interventions: Other: Traditional monitoring

INTERVENTIONS:
Device: WIN @ Hospital system — WIN @ Hospital system is a wearable and wireless system (Medical Class IIA) that allows continuous and real-time vital signs monitoring, automatically calculating the NEWS score with a personalized alert system for the patient. It does not require the continuous presence of the nurse in front of the control room, but is working with alert on portable devices (ipad).
  Arms: Vital signs wireless monitoring system
Other: Traditional monitoring — Vital signs control performed by nurse staff each 6 hours or more, according to medical advice.
  Arms: Control arm

SUMMARY:
The present study was planned to provide clinical data on the impact of acute and critically ill patients in Internal Medicine Unit activity and economic data enabling to quantify the relative cost of acute patients management during ordinary hospitalization. In these critically ill complex patients the vital parameters continuous monitoring could help in improving the quality of care. Therefore, the study will check how the wireless continuous monitoring in acute selected patients is able to reduce major complications improving the patient's outcome and the quality of care and reducing costs compared to traditional monitoring performed at regular intervals by the nursing staff.

DETAILED DESCRIPTION:
In recent years, Internal Medicine Ward, due to epidemiological transition, takes in charge more and more an heterogeneous group of patients with serious diseases both acute and chronic and elderly, frail, poly-pathological patients, requiring intensive care. Hospitalization of medical patients in large wards without prior stratification of severity, complexity, level of dependence, comorbidities and without a proper assessment of the risk of rapid clinical deterioration, can lead to suboptimal treatment, resulting in prolonged hospital stay and increased care costs. Continuous monitoring of vital parameters may allow early detection of deterioration in acute patients not admitted in intensive care such as those hospitalized in Internal Medicine Unit, allowing the staff to immediately address the patient's needs achieving promptly the most appropriate care. As there are no studies comparing the use of wireless monitoring systems and traditional vital signs monitoring in critical acute patients, the study was designed to highlight the benefits of continuous monitoring of vital signs in the first 72 hours hospitalization to reduce the major complications and improving outcome. The study also aims to assess the reduction in hospitalization costs using as proxy the decrease in average length of stay.

ELIGIBILITY:
Inclusion Criteria:

* all critical patients (with need for continuous monitoring and high technology) with MEWS ≥3 and / or NEWS≥5 at admission
* all patients with glycemic decompensation regardless of MEWS and NEWS.
* all critical patients severe fluid and electrolyte imbalance, regardless of MEWS and NEWS.

Exclusion Criteria:

* MEWS <3 and or NEWS <5
* Lack of informed consent
* Inability to understand and want

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2017-02-27 (Estimated); Primary Completion 2017-10-27 (Estimated); Study Completion 2018-02-27 (Estimated)

PRIMARY OUTCOMES:
Major complications reduction in subjects monitored with continuous wireless system | 12 months
  Reduction of major complications of critically ill patients from 15% to 5%.n subjects monitored with continuous wireless system

SECONDARY OUTCOMES:
Hospitalization costs reduction | 12 months
  1 day reduction of patient's average length of hospital stay

OTHER OUTCOMES:
Reduced nurse's time in monitoring vital parameters | 12 months
  Reduction of minutes of nursing commitment in monitoring vital parameters/ 24h
Patients' stratification according to level of intensity of care | 12 months
  Stratification of the patients hospitalized in Internal Medicine according to the level of intensity of care (using the MEWS score and NEWS - National Early Warning Scorei) and definition of end stage patients

CONTACTS AND LOCATIONS:
Overall Officials: Filomena Pietrantonio, MD, Principal Investigator — ASST GARDA
Locations (1):
- ASST-Garda Manerbio Hospital Internal Medicine Unit, Manerbio, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pietrantonio F, Orlandini F, Moriconi L, La Regina M. Acute Complex Care Model: An organizational approach for the medical care of hospitalized acute complex patients. Eur J Intern Med. 2015 Dec;26(10):759-65. doi: 10.1016/j.ejim.2015.08.011. Epub 2015 Sep 11. PMID 26365373
- [Background] Pietrantonio F, Scotti E. Internal medicine network: Is it a newsworthy idea? Eur J Intern Med. 2016 Nov;35:e18-e19. doi: 10.1016/j.ejim.2016.07.024. Epub 2016 Aug 4. No abstract available. PMID 27499176
- [Background] Vincent C, Amalberti R. Safer Healthcare: Strategies for the Real World [Internet]. Cham (CH): Springer; 2016. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK481869/ PMID 29465922
- [Background] Miglioramento della qualità della vita dei pazienti e riduzione del costo per il SSN attraverso l'uso di un sistema wireless di monitoraggio multi-parametrico dei parametri fisiologici. Case study sull'adozione del sistema di monitoraggio fisiologico WIN@Hospital presso l'Ospedale Campo di Marte, Lucca. Cangemi A, Turchetti B. Europe Health Summit Berlino (4-8 Maggio 2014)
- [Result] Pannick S, Wachter RM, Vincent C, Sevdalis N. Rethinking medical ward quality. BMJ. 2016 Oct 18;355:i5417. doi: 10.1136/bmj.i5417. No abstract available. PMID 27756729
- [Result] E. Scotti, F. Pietrantonio. The Hospital Internal Medicine Specialist today: a literature review and the SWOT analysis to elaborate a working proposal. Italian Journal of Medicine, vol 7, n.4 2013. 278-286. 1.08.2013
- [Result] F. Pietrantonio, L. Piasini, F. Spandonaro. Internal Medicine and emergency admissions: from a national Hospital Discharge Records (SDO) study to a regional analysis. . Italian Journal of Medicine Italian Journal of Medicine DOI: 10.4081/itjm.2016.674, vol 10, Issue 2, 2016
- [Result] Royal College of Physicians. National Early Warning Score (NEWS) Standardising the assessment of acute-illness severity in NHS. Report of a working party, July 2012.
- [Result] Orlandini F, Pietrantonio F, Moriconi L, La Regina M, Mazzone A, Campanini M. A model to improve the appropriateness in the management of acute poly-pathological patients: the acute complex care model http://dx.doi.org/10.4081/itjm.2016.697
- [Result] Subbe CP, Kruger M, Rutherford P, Gemmel L. Validation of a modified Early Warning Score in medical admissions. QJM. 2001 Oct;94(10):521-6. doi: 10.1093/qjmed/94.10.521. PMID 11588210
- [Result] Giovanna Bollini, Fabrizio Colombo. L'intensità assistenziale e la complessità clinica. Un progetto di ricerca della regione Lombardia. 2011
- [Result] Mongardi M, Bassi E, Di Ruscio E. Ospedale per Intensità di cura: strumenti per la classificazione dei pazienti. DGSPS, Servizio Presidi Ospedalieri, Regione Emilia-Romagna, Febbraio 2015
- [Result] Tartaglia R, Albolino S, Bellandi T, Bianchini E, Biggeri A, Fabbro G, Bevilacqua L, Dell'erba A, Privitera G, Sommella L. [Adverse events and preventable consequences: retrospective study in five large Italian hospitals]. Epidemiol Prev. 2012 May-Aug;36(3-4):151-61. Italian. PMID 22828228
- [Result] Charles V. Sicurezza del paziente. Edizione italiana a cura di Tartaglia R, Albolino S, Bellandi T. Milano, Springer-Verlag Italia, 2012.
- [Result] Institute of Medicine (US) Committee on Quality of Health Care in America; Kohn LT, Corrigan JM, Donaldson MS, editors. To Err is Human: Building a Safer Health System. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK225182/ PMID 25077248
- [Result] Bellocco A. Risk management in ospedale. Risk News CINEAS (Consorzio Universitario per l'Ingegneria nelle Assicurazioni) 2002;23.
- [Result] Programma Integrato di Miglioramento dell'Organizzazione (PIMO, Deliberazione N° X / 3652 Seduta del 05/06/2015)
- [Result] Sensium Science MF06-01, April 2015
- See also: Moher D, Hopewell S, Shulz KF, et al . The CONSORT statement: revised reccomendations for improving the quality of reports of parallel-group randomized trials.Evidence 2012; 4 (7): e1000024 www.consort-statement.org — http://www.consort-statement.org